CLINICAL TRIAL: NCT01718795
Title: Prehospital Laryngeal Tube vs. Bag-Valve Mask Ventilation Used by Paramedics During CPR- A Prospective, Controlled, Randomised, Multi-center Trial
Brief Title: Prehospital Laryngeal Tube vs. Bag-Valve Mask Ventilation Used by Paramedics During CPR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruiting too slow, down to 1-0 patients per month
Sponsor: Michael Baubin, MD (Other)
Responsible Party: Sponsor-Investigator, Michael Baubin, MD, Prof. MD, Medical University Innsbruck
Organization: Medical University Innsbruck (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prehospital LTS vs. BVM
Record Dates: First submitted 2012-06-07; First posted 2012-10-31 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Cardiac Arrest During and/or Resulting From A Procedure
Keywords: Airway; Cardiac Arrest; CPR; Ventilation
MeSH Terms: conditions — Heart Arrest; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bag-valve mask ventilation (Active Comparator): Bag-valve mask ventilation during CPR, i.e. traditional ventilation during CPR. Airway management with bag-valve mask ventilation and efficient ventilation: yes or no?
  Intervention is "Bag-valve mask ventilation" during CPR
  Interventions: Device: Bag-valve mask or laryngeal tube ventilation
- Laryngeal Tube (Active Comparator): Laryngeal Tube Ventilation during CPR, i.e. the alternative ventilation technique to be compared to the traditional technique. Airway management with laryngeal tube and efficient ventilation: yes or no?
  Intervention is "Ventilation through laryngeal tube" during CPR
  Interventions: Device: Bag-valve mask or laryngeal tube ventilation

INTERVENTIONS:
Device: Bag-valve mask or laryngeal tube ventilation — Interventions are either "Bag-valve mask (BVM)" or "Laryngeal tube (LT)" ventilation during CPR
  Other Names: BVM(Ambu,Germany);LT(VBM Medizintechnik,Germany)ventilation

SUMMARY:
During CPR bag-valve mask ventilation is difficult for basically skilled rescuers. Ventilation may be inefficient or with too high pressures result in stomach inflation and aspiration. Studies suggest that with a supraglottic airway device, such as the laryngeal tube, a basically skilled rescuer may ventilate more efficient and also safer. No prehospital study has been conducted comparing laryngeal tube and bag-valve mask ventilation during CPR. Thus, this study intends to compare ventilation with laryngeal tube and bag-valve mask performed by paramedics during CPR.

DETAILED DESCRIPTION:
During CPR bag-valve mask ventilation is difficult for basically skilled rescuers. Ventilation may be inefficient or with too high pressures result in stomach inflation and aspiration. Studies suggest that with a supraglottic airway device, such as the laryngeal tube, a basically skilled rescuer may ventilate more efficient and also safer. No prehospital study has been conducted comparing laryngeal tube and bag-valve mask ventilation during CPR. This study intends to compare ventilation with laryngeal tube and bag-valve mask performed by paramedics during CPR. This study may provide information if paramedics in an emergency should ventilate as they do traditionally with bag-valve mask ventilation or if they should ventilate with a laryngeal tube.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac arrest

Exclusion Criteria:

* Paramedic does not want to use laryngeal tube
* Physician on site before paramedic
* Foreign body airway obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2012-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Efficient ventilation | From start of paramedic ventilating the patient during CPR until emergency physician takes over ventilation or patient breathes again spontaneously after return of spontaneous circulation (ROSC)
  Does chest rise clearly during CPR? Thus efficient ventilation will be assessed during CPR, which may last on average between 20 and 60min. Therefore efficient ventilation will be assessed from starting CPR at 0min to 20min or rarely 60min or longer.

SECONDARY OUTCOMES:
Aspiration | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 month after enrollment of the last patient at August 30th 2014
  Aspiration will be assessed 24hrs after CPR with bronchoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Michael Baubin, Prof. MD, Principal Investigator — Medical University Innsbruck
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Fiala A, Lederer W, Neumayr A, Egger T, Neururer S, Toferer E, Baubin M, Paal P. EMT-led laryngeal tube vs. face-mask ventilation during cardiopulmonary resuscitation - a multicenter prospective randomized trial. Scand J Trauma Resusc Emerg Med. 2017 Oct 26;25(1):104. doi: 10.1186/s13049-017-0446-1. PMID 29073915
- See also: Departement of Anesthesiology and Critical Care Medicine Innsbruck, where study investigators belong to — http://www2.i-med.ac.at/anaesthesie/